CLINICAL TRIAL: NCT00687648
Title: Randomised Phase II Study of Metronomic Chemotherapy Plus the Same Aromatase Inhibitor Compared to Metronomic Chemotherapy Alone in Women With Hormone Receptor Positive, Her-2 Non-Overexpressing Advanced Breast Cancer Whose Disease Has Progressed While Receiving an Aromatase Inhibitor, Correlating Response With Circulating Endothelial Progenitor Cells, VEGF and VEGFR
Brief Title: Cyclophosphamide, Methotrexate, and Prednisolone With or Without Aromatase Inhibitor Therapy in Treating Postmenopausal Women With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000595712; SINGAPORE-NCC0706
Record Dates: First submitted 2008-05-30; First posted 2008-06-02 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; HER2-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Cyclophosphamide; exemestane; Letrozole; Methotrexate; Prednisolone

ARMS (2):
- Arm I (Experimental): Patients receive aromatase inhibitor (anastrozole, letrozole, or exemestane) as previously prescribed. Patients also receive oral cyclophosphamide once daily on days 1-28 and oral methotrexate twice on days 15, 16, 22, and 23 of course 1. For all subsequent courses, patients receive oral cyclophosphamide once daily and oral prednisolone once daily on days 1-28 and oral methotrexate twice on days 1, 2, 8, 9, 15, 16, 22, and 23. Treatment with cyclophosphamide, methotrexate, and prednisolone repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: anastrozole; Drug: cyclophosphamide; Drug: exemestane; Drug: letrozole; Drug: methotrexate; Drug: prednisolone
- Arm II (Active Comparator): Patients receive cyclophosphamide, methotrexate, and prednisolone as in arm I.
  Interventions: Drug: cyclophosphamide; Drug: methotrexate; Drug: prednisolone

INTERVENTIONS:
Drug: anastrozole — Given as previously prescribed
  Arms: Arm I
Drug: cyclophosphamide — Given by mouth
Drug: exemestane — Given as previously prescribed
  Arms: Arm I
Drug: letrozole — Given as previously prescribed
  Arms: Arm I
Drug: methotrexate — Given by mouth
Drug: prednisolone — Given by mouth

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, methotrexate, and prednisolone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Estrogen can cause the growth of breast cancer cells. Hormone therapy using anastrozole, letrozole, or exemestane may fight breast cancer by lowering the amount of estrogen the body makes. It is not yet known whether giving combination chemotherapy together with aromatase inhibitor therapy is more effective than combination chemotherapy alone in treating breast cancer.

PURPOSE: This randomized phase II trial is studying giving cyclophosphamide, methotrexate, and prednisolone together with aromatase inhibitor therapy to see how well it works compared with cyclophosphamide, methotrexate, and prednisolone in treating postmenopausal women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the clinical benefit rate (complete response, partial response or stable disease for > 24 weeks) in postmenopausal women with metastatic breast cancer treated with metronomic chemotherapy with vs without aromatase inhibitor therapy.

Secondary

* Compare the time to progression in these patients
* Compare the overall survival of these patients.
* Compare the safety and toxicity of these regimens in these patients.
* Correlate tumor response with markers of angiogenesis (circulating endothelial progenitor cells, VEGF, VEGF-C, VEGFR-2, and VEGFR-3).
* Determine the relative contribution of methotrexate and prednisolone to metronomic chemotherapy as assessed by change in circulating endothelial progenitor cell, VEGF, and VEGFR levels during serial addition of each drug.

OUTLINE: Patients are stratified according to site of metastases (visceral vs non-visceral only) and number of lines of prior chemotherapy in the metastatic setting (0 vs 1-2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive aromatase inhibitor (anastrozole, letrozole, or exemestane) as previously prescribed. Patients also receive oral cyclophosphamide once daily on days 1-28 and oral methotrexate twice on days 15, 16, 22, and 23 of course 1. For all subsequent courses, patients receive oral cyclophosphamide once daily and oral prednisolone once daily on days 1-28 and oral methotrexate twice on days 1, 2, 8, 9, 15, 16, 22, and 23. Treatment with cyclophosphamide, methotrexate, and prednisolone repeats every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive cyclophosphamide, methotrexate, and prednisolone as in arm I.

Patients undergo blood sample collection at baseline, in weeks 2, 4, 6, and 10, every 4 weeks until disease progression, and then at 4 weeks after disease progression. Blood samples are assessed for circulating endothelial progenitor cell levels by flow cytometry and VEGF, VEGF-C, VEGFR-2, and VEGFR-3 levels by ELISA immunoassays.

After completion of study therapy, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Metastatic disease
* Measurable disease, as defined by RECIST criteria
* Evidence of disease progression while receiving a third-generation aromatase inhibitor
* No extensive visceral disease (> 50% liver or lung parenchymal involvement)
* No pleural effusion or ascites
* No HER2/neu overexpression
* Hormone receptor status:

  * Estrogen receptor- or progesterone receptor-positive tumor

PATIENT CHARACTERISTICS:

* Postmenopausal, as defined by any of the following:

  * Over 60 years of age
  * 50-59 years of age with plasma follicle-stimulating hormone, luteinizing hormone, and estradiol in the postmenopausal range and amenorrhea for > 1 year
  * Any age with documented bilateral oophorectomy
* ECOG performance status (PS) 0-2 (Karnofsky PS 60-100%)
* Life expectancy > 6 months
* Leukocytes ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Total bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant
* Fertile patients must use effective contraception
* No other prior malignancies except curatively treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide, methotrexate, prednisolone, anastrozole, letrozole, or exemestane
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* No more than 2 lines of prior chemotherapy or endocrine therapy for advanced disease
* No other concurrent chemotherapy, immunotherapy, anticancer hormonal therapy, or anticancer surgery
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* No concurrent combination anti-retroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit response rate (complete response, partial response, or stable disease for > 24 weeks)

SECONDARY OUTCOMES:
Time to progression
Overall survival
Safety and toxicity
Correlation between tumor response and markers of angiogenesis
Relative contribution of methotrexate and prednisolone to metronomic chemotherapy as assessed by change in circulating endothelial progenitor cell, VEGF, and VEGFR levels during serial addition of each drug

CONTACTS AND LOCATIONS:
Overall Officials: Wong Nan Soon, MBBS, MRCP, FAMS, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre - Singapore, Singapore, Singapore